CLINICAL TRIAL: NCT03620877
Title: A Program for Improved Family Screening for Colorectal Cancer
Acronym: COLOR3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: COLOR 3
Record Dates: First submitted 2018-06-21; First posted 2018-08-08 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- personalized intervention (Experimental): Personalized intervention by a preventive nurse, relying on validated prevention models, in improving participation in the colonoscopic screening of siblings
  Interventions: Behavioral: Personalized intervention

INTERVENTIONS:
Behavioral: Personalized intervention — Personalized intervention by a preventive nurse, relying on validated prevention models, in improving participation in the colonoscopic screening of siblings

SUMMARY:
A first- degree family history of colorectal cancer (CRC) or adenoma before age 65 is associated with a high risk of CRC. For these high-risk subjects, the French 2013 recommendations advise colonoscopy screening, but participation is insufficient (26-54%).The purpose of this project is to propose, through association of multidisciplinary research teams (public health, sociology, linguistic), actors on the field (physicians, organized screening facilities), and decision makers, relevant and effective interventions in the framework of a public health program, enabling increased participation of relatives of patients with CRC or adenoma before age 65 in targeted screening for CRC by colonoscopy.

DETAILED DESCRIPTION:
A first-degree family history of colorectal cancer (CRC) or adenoma before age 65 is associated with a high risk of CRC. For these high-risk subjects, the French 2013 recommendations advise colonoscopy screening, but participation is insufficient (26-54%).The purpose of this project is to propose, through association of multidisciplinary research teams (public health, sociology, linguistic), actors on the field (physicians, organized screening facilities), and decision makers, relevant and effective interventions in the framework of a public health program, enabling increased participation of relatives of patients with CRC or adenoma before age 65 in targeted screening for CRC by colonoscopy.

Description of the intervention: This program, offered in 4 departments is divided into 3 phases:

1. Sensitization of doctors to the recommendations. This is a collaborative work with clinicians to enable them i) to take ownership of the problem and generic documents used in the previous study and ii) to define an intervention logic to encourage them to systematically inform subjects with RCC or advanced adenoma before age 65 the increased risk related to their 1st degree.
2. Coordinated transmission of information from the patient's physician to the relative's physician under consent of the patient and his/her relatives. Under the terms established with the actors in the previous phase, the physician delivers standard information to the index patient, presents the generic documents and may adapt the procedure to each patient's needs. With support of the coordination team which collects the coordinates of 1st degree relatives, the patient's physician transmits the information to the relatives and their doctors. The coordination team, during this experimental phase, will be the team of Epidemiology, Cancer Registry of Poitiers University Hospital, under the responsibility of public health physicians. The coordination team contacts each relative on behalf of the index patient's consent, acting by delegation of the index patient's physician, informs about the transmission of information given to the index patient, requests the agreement of the relative that the patient's doctor would contact his/her doctor to inform, under cover of professional secrecy, of the medical context.
3. Personalized information of relatives by a preventive nurse based on validated prevention models (individual psychosocial factors associated with screening and behavioral stage). At most two years after diagnosis of the index patient, the relative's colonoscopy performance status will be ascertained by the coordination team in connection with the attending physician. If the relative has had a colonoscopy carried out, the coordination team shall document the results and note the date scheduled for the following exam. If the relative has not had a colonoscopy carried out, he shall then receive a personalized intervention, based on the intervention evaluated in the previous study, as a supplement to the action of his/her doctor.

Qualitative and quantitative evaluations will follow each phase to measure the acceptability, coverage, efficiency, to assess transferability of the program. Moreover the program will be evaluated by a population survey conducted by the cancer registry that covers the geographical area of the experimentation with data collection that identify exhaustively the patients with CRC or high-grade adenoma.

ELIGIBILITY:
Inclusion Criteria:

* First-degree relatives of an index patient: father, mother, children, brothers and sisters (aged more than 18 years).

Informed and oral consent of the participant after clear and fair information on the study

Exclusion Criteria:

* The persons concerned by the articles L.1121-5 to L1121-8 and L.1122-1-2 of the Code de la santé publique will not be included in the interviews of the qualitative studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of coordinated transmission | 18 months
  Colonoscopies carried out by relatives

SECONDARY OUTCOMES:
Evaluation of doctors' sensitization to the recommendations. | up to 10 months
  Group interviews with physicians to bring together their opinions and to validate the program modalities
Adherence to personalized intervention | 24 months
  On-telephone and face-to-face interviews with physicians and relatives.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Ingrand, MD, PhD, Study Director — University Hospital, Poitiers, France
Locations (1):
- INGRAND, Poitiers, France

REFERENCES:
- [Background] Butterworth AS, Higgins JP, Pharoah P. Relative and absolute risk of colorectal cancer for individuals with a family history: a meta-analysis. Eur J Cancer. 2006 Jan;42(2):216-27. doi: 10.1016/j.ejca.2005.09.023. Epub 2005 Dec 9. PMID 16338133
- [Background] Ingrand I, Defossez G, Richer JP, Tougeron D, Palierne N, Letard JC, Beauchant M, Ingrand P. Colonoscopy uptake for high-risk individuals with a family history of colorectal neoplasia: A multicenter, randomized trial of tailored counseling versus standard information. Medicine (Baltimore). 2016 Aug;95(33):e4303. doi: 10.1097/MD.0000000000004303. PMID 27537555
- [Background] Taouqi M, Ingrand I, Beauchant M, Migeot V, Ingrand P. Determinants of participation in colonoscopic screening by siblings of colorectal cancer patients in France. BMC Cancer. 2010 Jul 6;10:355. doi: 10.1186/1471-2407-10-355. PMID 20602807
- [Background] Ingrand I, Dujoncquoy S, Beauchant M, Letard JC, Migeot V, Ingrand P. General practitioner and specialist views on colonoscopic screening of first-degree relatives of colorectal cancer patients. Cancer Epidemiol. 2009 Oct;33(3-4):223-30. doi: 10.1016/j.canep.2009.07.002. Epub 2009 Aug 3. PMID 19683486
- [Background] Ingrand I, Dujoncquoy S, Migeot V, Ghadi V, Beauchant M, Ingrand P. Interactions among physicians, patients, and first-degree relatives in the familial screening of colorectal cancer in France. Patient Prefer Adherence. 2008 Feb 2;2:47-55. PMID 19920944
- [Background] Ng SC, Lau JY, Chan FK, Suen BY, Tse YK, Hui AJ, Leung-Ki EL, Ching JY, Chan AW, Wong MC, Ng SS, To KF, Wu JC, Sung JJ. Risk of Advanced Adenomas in Siblings of Individuals With Advanced Adenomas: A Cross-Sectional Study. Gastroenterology. 2016 Mar;150(3):608-16; quiz e16-7. doi: 10.1053/j.gastro.2015.11.003. Epub 2015 Nov 14. PMID 26584600